CLINICAL TRIAL: NCT06452901
Title: PROgressive struCturEd Simulation-based Surgical Training Program (PROCESS) - Open Vascular Surgery
Acronym: PROCESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Responsible Party: Principal Investigator, Camilo Alejandro Velandia Sánchez, Mandatory Social Service Medical Doctor, Fundación Cardioinfantil Instituto de Cardiología
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEIC-013-2024
Record Dates: First submitted 2024-05-20; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Vascular Diseases; Competency-Based Education; Simulation Training
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: A triple-arm, randomized, simple-blinded clinical trial will be conducted. A control sequence and an intervention sequence of three subgroups with different exposure levels to the simulation program are proposed. Group 1: open abdominal aortic repair (AAOR), Group 2: vascular anastomosis (VA) and AAOR, and Group 3: specific micro-surgical skills, VA and AAOR
Who Masked: Outcomes Assessor
Masking Description: Evaluators, who are external to the researchers, will be single-blinded to assess the effectiveness of different interventions. They will remain unaware of the participants' group assignments. Privacy will be maintained through coding and presenting de-identified data. Data will also be presented without voices, glove usage, and image distortion to prevent identification of personal details such as gender, race, or other characteristics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Will receive the complete structured and progressive training program involving specific micro-surgical skills, VA, and AAOR.
  Interventions: Other: Progression and structured surgical training.
- Group II (Active Comparator): Will only receive VA and AAOR training.
  Interventions: Other: Progression and structured surgical training.
- Group III (Active Comparator): Will only receive AAOR training.
  Interventions: Other: Progression and structured surgical training.

INTERVENTIONS:
Other: Progression and structured surgical training. — Participants will be exposed to different amounts of open vascular surgical training, but only group I will receive the complete structured and progressive training program. This ensures that all participants have access to the potential benefits derived from the intervention. Current evidence supports this approach, which supports the benefits of medical simulation in the training process of surgical residents.

SUMMARY:
A triple-arm, randomized, simple-blinded clinical trial will be conducted. A control sequence and an intervention sequence of three subgroups with different exposure levels to the simulation program are proposed. Group 1: open abdominal aortic repair (AAOR), Group 2: vascular anastomosis (VA) and AAOR, and Group 3: specific micro-surgical skills, VA and AAOR. Surgical residents of general, vascular, or cardiovascular surgery programs will be included. Sample size calculation resulted in 45 participants, 15 in each group. Simple blinding will involve external evaluators. Randomization will occur as a simple randomization.

ELIGIBILITY:
Inclusion Criteria:

* Vascular Surgery, Cardiothoracic Surgery, and General Surgery residents.
* Over 18 years old.

Exclusion Criteria:

* Serious illnesses, such as advanced cancer, decompensated cardiovascular diseases, or severe neurological disorders, could be exclusion criteria due to concerns about the participant's safety and ability to complete the study.
* Participants who have known allergies to components of the interventions or have experienced severe adverse reactions in the past will be excluded from the study.
* Any medical condition that could interfere with the participant's ability to complete assessments or follow study guidelines could be a reason for exclusion. This could include, for example, severe physical disabilities or illnesses requiring continuous hospitalization.
* Individuals who cannot provide valid informed consent due to cognitive issues, mental impairment, or legal incapacity will be excluded from the study.
* Individuals who have had prior exposure to structured simulation programs in vascular surgery will be excluded. Previous familiarity with simulation could influence study outcomes, introducing a prior learning bias that could distort the assessment of the intervention's effectiveness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-21 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy in the acquisition of technical surgical skills. | 4 months
  Pre- and post-intervention individual measures will be taken using the OPEn Aortic Aneurysm Repair Assessment of Technical Expertise (OPERATE) tool to compare the efficacy of the simulated program. The unit of measure are the points of OPERATE Scale with a established passing score of 27.7. A higher score means a better outcome.

SECONDARY OUTCOMES:
The efficacy given by the progression through the different structured modules. | 4 months
  The results of the 3 arms will be compared. The unit of measure are the points of OPERATE Scale with a established passing score of 27.7. A higher score means a better outcome.
The satisfaction of the residents | 4 months
  Surveys guided by a Likert Scale will measure the Level 1 of Kirkpatricks levels based on the reaction and satisfaction of the participants after the implementation of the interventions.
  The unit of measure will be the result on the Likert scale; the minimum score is 1, and the maximum is 10. A higher score means a better outcome.

IPD SHARING:
Plan to Share IPD: No
The data may not be available for public access due to participant privacy concerns but may be available from the corresponding author upon reasonable request.